CLINICAL TRIAL: NCT01722175
Title: Associating Liver Partition With Portal Vein Ligation for Staged Hepatectomy (ALPPS) Versus Portal Vein Occlusion (PVO) to Induce Liver Regeneration for Resection of Liver Tumors That Are Unresectable in One Step - a Randomized Controlled Trial
Brief Title: Associating Liver Partition With Portal Vein Ligation For Staged Hepatectomy (ALPPS) or Portal Vein Occlusion in Treating Patients With Liver Cancer
Acronym: ALPPS
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Safety concerns.
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201209123
Record Dates: First submitted 2012-11-02; First posted 2012-11-06 (Estimated); Last update posted 2014-07-22 (Estimated); Status verified 2014-07

CONDITIONS: Carcinoma, Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (ALPPS) (Experimental): Patients undergo Associating Liver Partition with Portal Vein Ligation (ALPPS) step 1 surgery on day 0 and step 2 surgery 7-14 days later, based on patient's liver size.
  Interventions: Procedure: ALPPS surgery
- Arm II (PVO) (Active Comparator): Patients undergo portal vein occlusion (PVO) step 1 on day 0 and step 2 surgery 6-8 weeks later, based on patient's liver size.
  Interventions: Procedure: PVO surgery

INTERVENTIONS:
Procedure: ALPPS surgery
  Arms: Arm I (ALPPS)
Procedure: PVO surgery
  Arms: Arm II (PVO)

SUMMARY:
This randomized phase II trial compares how well associating liver partition with portal vein ligation for staged hepatectomy (ALPPS) or portal vein occlusion (PVO) works in treating patients with liver cancer. Both treatments are types of 2-stage hepatectomies for removing liver cancer. ALPPS may be more effective than PVO in patients whose disease would traditionally be considered inoperable.

ELIGIBILITY:
Inclusion Criteria:

* Patient may have primary or secondary hepatic malignancies with a FLR/TLV < 30% or a FLR/BW ratio of < 0.5 for patients with normal liver function (defined as normal transaminases, normal bilirubin, normal factor V, and normal PT/INR). In case of injury due to chemotherapy, known high grade steatosis, or cholestasis > 50 mmol/L, patient may be enrolled into the trial if FLR/TLV is < 40% or FLR/BW ratio < 0.8.
* Patient must have extensive liver tumors that would require portal vein embolization or a two-stage hepatectomy and portal vein embolization or ligation by the judgment of surgeons in the tumor board.
* Patient may have extrahepatic disease as long as it may be addressed after liver surgery and there is a tumor board decision to proceed with liver resection (mostly applicable to CRC metastases).
* Patient may have received previous chemotherapy.
* In cases of cholestasis, preoperative drainage procedures (PTC or ERCP) are left up to judgement of physicians.
* Patient must be ≥ 18 years of age. The patient population over 65 years old needs to be carefully included based on comorbidities.
* Patient may have undergone previous liver resection.
* Patient's location must be such that proper staging and follow-up may be performed.
* Patient's case must be presented at the Multidisciplinary Meeting attended by hepatobiliary surgeons, oncologists, hepatologists, and radiologists, or must be approved directly by Dr. Strasberg or Dr. Chapman.
* Patient must be able to understand and willing to sign a written informed consent document.

Exclusion Criteria:

* Patient must not have any significant concomitant diseases rendering him/her unsuitable for major liver surgery by the judgment of the physicians involved, especially if the patient is > 65 years old.
* Patient must not have enrolled into a clinical trial within 4 weeks of study entry.
* Patient must not have peritoneal carcinomatosis or other extensive extrahepatic disease.
* Patient must not have advanced stages of carcinoma of the gallbladder (T3/T4)
* Patient must not have issues such as drug and/or alcohol abuse.
* Patient must not need major extrahepatic surgery (e.g. pancreas resection, gastric resection, rectal surgery) within 3 months of study entry.
* Patient must not be a candidate for liver transplantation in case of HCC.
* Patient must not be pregnant or breastfeeding. If a female of childbearing potential, patient must have a negative pregnancy test within 14 days of enrollment.

Inclusion of Women and Minorities

-Both men and women and members of all races and ethnic groups are eligible for this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2016-04 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Liver free of tumors | At 3 months
  Assessed by two independent and blinded radiologists using dynamic MRI with liver specific contrast; proportion of patients in each treatment arm; incidence across two arms will be summarized using contingency tables and compared by 2-sample Chi-square test or Fisher's exact test.

SECONDARY OUTCOMES:
Overall survival | Up to 3 years
  Kaplan-Meier product limit estimator will be used to describe the distribution of overall survival (OS). The differences in OS between treatment arms will be compared using log-rank test.
Disease-free survival | Up to 3 years
  Kaplan-Meier product limit estimator will be used to describe the distribution disease-free survival (DFS). The differences in DFS between treatment arms will be compared using log-rank test.
Incidence of complications | 3 months
  Each patient will be categorized according to the most severe complication occurring during the two procedures of each arm; distributions across two arms will be compared by 2-sample Chi-square test or Fisher's exact test.
Liver volumetric change after step 1 of ALPPS or PVO | 8 weeks
  Assessed at 1, 2, 4 and 8 weeks after step 1 using CT or MRI imaging; differences between two arms will be compared using 2-way ANOVA for repeated measurement data
Liver synthetic and transport function | 3 months
  PT/INR, factor V and bilirumen are measured; differences between two treatment arms will be compared using t-test or Mann-Whitney rank-sum test as appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Strasberg, M.D., Principal Investigator — Washington University School of Medicine

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu